CLINICAL TRIAL: NCT05285670
Title: Mobile Solutions to Empower Reproductive Life Planning for Women Living With HIV
Brief Title: Mobile Phone Messaging to Improve Reproductive Health for Women Living With HIV in Kenya (Mobile WACh Empower)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Alison Drake, Associate Professor, SPH: Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00013136; R01HD104551 (NIH)
Record Dates: First submitted 2022-02-18; First posted 2022-03-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hiv; Contraception; Fertility Issues
Keywords: mHealth; HIV; conception; counseling; fertility; family planning; SMS; Kenya
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infertility

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to 1) A digital counseling tool plus interactive two-way SMS dialogue or 2) Control (no SMS) at the clinic level, using 1:1 allocation at the clinic level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital counseling plus interactive two-way SMS dialogue (Experimental): Participants will receive initial counseling on a tablet followed by automated SMS messages with prompts to reply. They will have the ability to both respond to and initiate SMS dialogue. Trained Study Nurses will monitor and respond to participant messages.
  Interventions: Behavioral: Digital counseling plus interactive two-way SMS dialogue
- Control (No Intervention): Control receiving standard of care.

INTERVENTIONS:
Behavioral: Digital counseling plus interactive two-way SMS dialogue — We will utilize a digital counseling tool on a tablet to provide initial reproductive life planning counseling while waiting for an HIV care provider. We will then use Mobile WACh, a human-computer hybrid system that enables seamless two-way SMS communication and patient tracking, to provide consistent support to women following enrollment and for up to 2 years. Women will receive automated theoretically grounded SMS messages targeting the appropriate reproductive health needs and will have the capability to respond and spontaneously message a nurse based at the clinic. . Automated SMS will be delivered at times and in languages based on patient preferences, weekly the first 3 months, every other week in months 4-12, and monthly during the last year of the trial. If there is a change in the reproductive health needs, more frequent messaging will be re-initiated at the same frequency as enrollment.
  Arms: Digital counseling plus interactive two-way SMS dialogue

SUMMARY:
Use of a mobile health (mHealth) intervention to provide reproductive life counseling to women living with HIV may improve delivery of integrated reproductive health/HIV services and prevent adverse reproductive health outcomes. The proposed study will evaluate SMS platform and reproductive health counseling intervention in a cluster randomized controlled trial among women receiving routine HIV care, and plan for future implementation with qualitative and health economic analyses.

DETAILED DESCRIPTION:
Meeting reproductive health needs of women living with HIV (WLWH) is essential to help women prevent unintended pregnancies, safely conceive, and eliminate mother-to-child HIV transmission (MTCT). Reproductive life planning is complex for WLWH, who are faced with making decisions about antiretroviral treatment selections and potential for drug interactions with contraceptive methods, planning for safe conception, and planning to prevent sexually transmitted infections. While family planning (FP) use is high among WLWH, discontinuation of FP is common among women who desire pregnancy prevention, and is an important driver of unmet need for FP and subsequent risk of unintended pregnancy and adverse maternal and child health outcomes. Many programs in sub-Saharan Africa integrate FP service delivery into routine HIV care, but HIV care providers face challenges with implementing these models of care. HIV care providers may be ill equipped to ensure WLWH receive high-quality, rights' based reproductive health counseling and services due to lack time, training, resources, and skills. Prior studies on integrating FP services into HIV care consistently cite implementation challenges. Mobile health technology may provide a low cost solution to augment counseling services, strengthen health care systems, and alleviate demands on HIV providers. The investigators hypothesize that providing comprehensive counseling and two-way SMS communication, will 1) improve delivery of integrated HIV and reproductive health care services, 2) reduce contraceptive discontinuation rates, 3) be acceptable and feasible to implement, and 4) be cost-effective and contribute to prevention MTCT efforts. The investigators will adapt a unique two-way SMS platform (Mobile WACh) that combines automated bulk SMS messaging and dialogue with a health care provider for a new population, new environment, and new outcomes for long-term impact. The Mobile WACh platform will be customized to provide continuous reproductive life planning counseling for WLWH. The investigators will test the combined intervention in a cluster randomized controlled trial among women receiving HIV care at 10 facilities in Kenya (330 per facility). The investigators propose to evaluate the effect of the counseling and SMS communication intervention, Mobile WACh Empower, on reproductive health outcomes. In Aim 1, the investigators will determine the effect of the Mobile WACh Empower intervention on FP discontinuation, dual method use, and unmet need for FP over 2 years. In Aim 2, the investigators will evaluate acceptability, feasibility, and scalability of implementing Mobile WACh Empower under real-world settings, from both WLWH and provider perspectives in focus group discussions. In Aim 3, the investigators will construct a mathematical model to measure health and economic impacts of Mobile WACh Empower, including cost-effectiveness of the intervention per pregnancy and MTCT averted. This trial will evaluate a novel intervention to address a crucial gap in provision of integrated reproductive health and HIV care, and has the potential to make a significant contribution to global goals of universal access to FP and elimination of MTCT.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Receiving HIV care at study site
* Reproductive age (18-45; 14-17 if emancipated minors)
* Daily access to mobile phone (own phone or shared)
* Plan to receive HIV care at enrollment facility for 2 years
* Speak English, Kiswahili, or Luo
* Literate or comfortable with someone reading study SMS

Exclusion Criteria:

* Currently pregnant

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3310 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Contraceptive discontinuation | 2 years
  Proportion not using contraception among women who initiated or continued contraception to prevent pregnancy

SECONDARY OUTCOMES:
Uptake of dual methods of contraception | 2 years
  Proportion who use condoms plus another modern method of contraception
Unmet need for contraception | 2 years
  Proportion with a desire for pregnancy but not using contraception

OTHER OUTCOMES:
Viral load suppression at conception | Up to 2 years
  Proportion with viral load <100 copies/mL among women planning to become pregnant or become pregnant
Unintended pregnancy | 2 years
  Proportion of women who become pregnant among women not intending pregnancy (excludes ambivalence)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Drake, PHD, Principal Investigator — University of Washington
Locations (10):
- Kenya (10):
  - Bondo sub-County Hospital, Bondo
  - Kisumu District General Hospital, Kisumu
  - Lumumba sub-County Hospital, Kisumu
  - Dandora 2 Health Center, Nairobi
  - Kangemi Health Centre, Nairobi
  - Kenyatta National Hospital, Nairobi
  - Mathare North Health Center, Nairobi
  - Riruta Health Center, Nairobi
  - Rachuonyo District, Oyugis
  - Siaya District Hospital, Siaya

IPD SHARING:
Plan to Share IPD: Yes
Data from Mobile WACh Empower will be available at end of the project by contacting the study team at the University of Washington. De-identified data and variables requested.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: At the end of the study, available for 5 years

REFERENCES:
- [Background] Ngumbau N, Unger JA, Wandika B, Atieno C, Beima-Sofie K, Dettinger J, Nzove E, Harrington EK, Karume AK, Osborn L, Sharma M, Richardson BA, Seth A, Udren J, Zanial N, Kinuthia J, Drake AL. Mobile solutions to Empower reproductive life planning for women living with HIV in Kenya (MWACh EMPOWER): Protocol for a cluster randomized controlled trial. PLoS One. 2024 Apr 1;19(4):e0300642. doi: 10.1371/journal.pone.0300642. eCollection 2024. PMID 38557692